CLINICAL TRIAL: NCT02071667
Title: Association of Periostin Levels and Chronic Sinusitis
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit/enroll subjects for study.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, John Steinke, Associate Professor, University of Virginia
Other Study IDs: 17123
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Sinusitis; Nasal Polyps
Keywords: Chronic sinusitis; Nasal Polyps
MeSH Terms: conditions — Sinusitis; Nasal Polyps | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and paraffin embedded nasal polyp tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects who require sinus surgery
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw

SUMMARY:
The purpose of this study is to see if a protein in blood, called periostin, can determine if patients have chronic sinusitis. This protein is in everyone's body, but the level of the protein may indicate certain conditions such as chronic sinusitis. The investigators are interested in testing levels of periostin to see if they are higher or lower than patients without chronic sinusitis, just as periostin is higher in patients with asthma. All patients enrolled in this study will have chronic sinusitis without asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sinus disease which requires surgical intervention
* Ability to understand and give informed consent

Exclusion Criteria:

* Previous diagnosis of asthma
* Positive methacholine challenge at screening
* Diagnosis of cystic fibrosis
* Concomitant use of systemic corticosteroids (except for those prescribed as part of standard pre-surgical treatment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are recommended for sinus surgery as part of their care who self report no asthma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Difference in circulating serum periostin levels pre and post sinus surgery | 10-15 weeks
  Serum collected prior to and following sinus surgery will be analyzed for concentrations of the protein periostin.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States